CLINICAL TRIAL: NCT03526367
Title: A Randomized Trial of Rosuvastatin Loading Combined With Early hydrAtion Versus Standard-of-care Medications for the Prevention of Contrast Induced Acute Kidney Injury in Patient With Acute Myocardial Infarction Undergoing Emergency Percutaneous Coronary Intervention (TRACK-AMI)
Brief Title: A Randomized Trial of Rosuvastatin Loading Combined With Early hydrAtion Versus Standard-of-care Medications for the Prevention of CIAKI in Patient With AMI Undergoing Emergency PCI
Acronym: TRACK-AMI
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study withdrawn for no sufficient fund support.
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Prof., Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TRACK-AMI V1.0
Record Dates: First submitted 2018-04-25; First posted 2018-05-16 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Contrast-induced Acute Kidney Injury; ST Elevation Myocardial Infarction; Primary PCI; Rosuvastatin; Hydration
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydration plus rosuvastatin therapy (Experimental): 1. After randomized，hydration（3ml/kg/h, if patients had LVEF<40%, 1.5 ml/kg/h）last 12 hours;
  2. After randomized，a loading dose of rosuvastatin 20mg then 10 mg daily followed for at least 7 days.
  Interventions: Drug: hydration plus rosuvastatin therapy
- Standard therapy (Active Comparator): No statin within 12 h after randomization, hydration at physicians' discretion, but no more than 1ml/kg/h.
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: hydration plus rosuvastatin therapy — In experimental group,a loading dose of rosuvastatin 20mg then 10 mg daily followed for at least 7 days and hydration（3ml/kg/h）last 12 hours after randomized
  Arms: hydration plus rosuvastatin therapy
Drug: Standard therapy — Prohibition of use any statins from randomized to 12 hours after procedure; The hydration or not is determined by physicians but 1 ml/kg/h at most.
  Arms: Standard therapy

SUMMARY:
The CIAKI,as the third complication of PCI, was associated with adverse cardiac events after procedure. Moreover, because the rate of periprocedure hydration is inadequate in STEMI patients before primary PCI, the incidence of CIAKI is higher significantly in these patients. The cardiovascular pleiotropic effects of statins in addition to lipid have been widely concerned. The previous studies demonstrated usage of statin in periprocedure could decrease the risk of CIAKI. Compared with hydration, the usage of statin to prevention CIAKI show the advantages in clinical practice, for example，there is no need to consider the cardiac function.The optimal strategies for preventting CIAKI in STEMI patients undergoing primary PCI needed further studies to explore. What's more, whether a synergistic effect of hydration and statin or not is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old
* The STEMI patients within 12 h of onset(or within 12-24 h of onset with chest pain and persistent ST-segment elevation or the presence of a new LBBB);
* The patients planned primary PCI;
* At least one of the following:

Diabetes mellitus, Chronic Kidney Disease, Female, Elder(Age≥65), Hypertension class 3, Congestive heart failure

• Voluntary signature of informed consent

Exclusion Criteria:

* Type 2 Myocardial infarction secondary to an ischaemic imbalance
* Intolerance of statin or iodine contrast
* eGFR<30ml/min
* Administration of any iodinated (e.g.CT angiography) within 14 days before enrollment
* Hepatic dysfunction, ALT 3 times greater than upper normal limit
* Thyreoid insufficiency
* Hemodynamic instability
* Have received PCI or CABG within 30 day before enrollment
* Plan to perform any coronary angiography or PCI within 30 days
* Have received any statins within 7 days before enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-20 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
CIAKI | 7 days
  CIAKI, defined an Absolute Increase in SCr ≥0.5mg/dL（≥44.2μmmol/L）or a ≥ 25% Increase in SCr From Baseline to 7 days After the Procedure

SECONDARY OUTCOMES:
The peak value of Scr | withtin 7 days before randomized
The rate of Aggravated Heart Function | withtin 30 days before randomized
  Aggravated at Least 1 Class of Heart Function
The rate of Hospitalization for Aggravated Renal Function, Acute Renal Failure, Dialysis or Hemofiltration | withtin 30 days before randomized
the level of hsCRP | withtin 7 days before randomized
The Composite of all-cause death, MI, stroke, and TVR | withtin 30 days before randomized

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Principal Investigator — The General Hospital of Shenyang Millitary Region
Locations (1):
- The General Hospital of Shenyang Millitary Region, Shenyang, Liaoning, China